CLINICAL TRIAL: NCT05398536
Title: Kinesiophobia and Related Factors in Adult Patients With Familial Mediterranean Fever
Brief Title: Kinesiophobia in Familial Mediterranean Fever
Status: Completed | Type: Observational
Sponsor: Halic University (Other)
Responsible Party: Principal Investigator, Seda Saka, PT PhD, Halic University
Other Study IDs: ssaka6
Record Dates: First submitted 2022-05-26; First posted 2022-06-01 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: FMF
Keywords: Kinesiophobia; fear-avoidance; physical activity; familial Mediterranean fever
MeSH Terms: conditions — Kinesiophobia; Motor Activity; Familial Mediterranean Fever

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Kinesiophobia is a common problem in patients with rheumatic disease and can cause physical inactivity, social isolation, disability, and poor quality of life. This study aimed to evaluate kinesiophobia and associated factors in patients with familial Mediterranean fever (FMF). All patients were evaluated in terms of sociodemographic characteristics and assessed using the Tampa Kinesiophobia Scale (TKS), International Physical Activity Questionnaire (IPAQ), Fatigue Severity Scale (FSS), and Hospital Anxiety and Depression Scale (HADS).

DETAILED DESCRIPTION:
Familial Mediterranean fever (FMF) is a common autoinflammatory disease among certain ethnic groups living in the Mediterranean basin. The reported prevalence of FMF among children in Turkey is 9.3/10000. Kinesiophobia is a common problem in patients with rheumatic disease and can cause physical inactivity, social isolation, disability, and poor quality of life. This study aimed to evaluate kinesiophobia and associated factors in patients with familial Mediterranean fever (FMF). All patients were evaluated in terms of sociodemographic characteristics and assessed using the Tampa Kinesiophobia Scale (TKS), International Physical Activity Questionnaire (IPAQ), Fatigue Severity Scale (FSS), and Hospital Anxiety and Depression Scale (HADS).

ELIGIBILITY:
Inclusion Criteria:

* being age over 18
* being volunteer

Exclusion Criteria:

* ortopedic, neurologic, cardiopulmonary diseases that prevent physical activity
* psychological diagnosis and drug usage

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The authors contacted the president of the national Behçet's Disease and Familial Mediterranean Fever Patients Association. The president invited members to participate in the study by e-mail.
Sampling Method: Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2018-01-08 (Actual); Primary Completion 2018-03-27 (Actual); Study Completion 2018-12-20 (Actual)

PRIMARY OUTCOMES:
Tampa Kinesiophobia Scale (TKS) | at the enrollment
  The TKS consists of 17 items scored on a 4-point Likert scale and measures fear of movement/(re)injury. The questions include the parameters of injury/reinjury and fear-avoidance in work-related activities [15]. The total score is obtained by summing all items, and a higher score indicates greater fear of movement. A total score greater than 37 is regarded as indicating a high level of kinesiophobia
Hospital Anxiety and Depression Scale (HADS) | at the enrollment
  The scale consists of 14 items divided into the depression and anxiety subscales, each with 7 items. The items on the scale are scored from 0 to 3 using a 4-point Likert scale. The scores of the odd-numbered items are summed to obtain the anxiety subscale (HADS-A) score and the even-numbered items are summed to obtain the depression subscale (HADS-D) score. Possible scores for each subscale range from 0 to 21.
International Physical Activity Questionnaire (IPAQ) | at the enrollment
  In the IPAQ, respondents estimate how often and for how long they engaged in various activities in the last 7 days. To determine PA levels, the known metabolic equivalent (MET) for each activity is multiplied by its duration and frequency to obtain a score in MET minutes. MET values used in this study were 8.0 for vigorous physical activity (VPA) [8, 19], 4.0 for moderate physical activity (MPA), and 3.3 for light physical activity (LPA). The overall PA score is calculated by summing the results of all items [20]. PA levels were classified into 3 categories: inactive (<600 MET-min/week), low PA level (600-3000 MET-min/week), and adequate PA level (>3000 MET-min/week)

CONTACTS AND LOCATIONS:
Overall Officials: Seda Saka, PT, PhD, Principal Investigator — Haliç University
Locations (1):
- Haliç University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Oskay D, Tuna Z, Duzgun I, Elbasan B, Yakut Y, Tufan A. Relationship between kinesiophobia and pain, quality of life, functional status, disease activity, mobility, and depression in patients with ankylosing spondylitis. Turk J Med Sci. 2017 Nov 13;47(5):1340-1347. doi: 10.3906/sag-1702-93. PMID 29151302
- [Result] Giese A, Ornek A, Kilic L, Kurucay M, Sendur SN, Lainka E, Henning BF. Anxiety and depression in adult patients with familial Mediterranean fever: a study comparing patients living in Germany and Turkey. Int J Rheum Dis. 2017 Dec;20(12):2093-2100. doi: 10.1111/1756-185X.12297. Epub 2014 Jan 28. PMID 24467729